CLINICAL TRIAL: NCT05478239
Title: Phase II Trial of ArtemiCoffee for Men With Biochemical Recurrence of Prostate Cancer After Initial Local Therapy
Brief Title: ArtemiCoffee in Patients With Rising PSA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zin W Myint (Other)
Collaborators: ArtemiLife (Unknown)
Responsible Party: Sponsor-Investigator, Zin W Myint, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22-GU-79
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Artemisia annua; Biochemically recurrent; Prostate-specific antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prostate cancer patients (Experimental): Men with biochemical recurrence of prostate cancer after initial local therapy.
  Interventions: Drug: ArtemiCoffee

INTERVENTIONS:
Drug: ArtemiCoffee — 3 cups of Artemisia annua (Aa) coffee per day (1350mg) for 24 weeks.
  Other Names: Artemisia annua (Aa) coffee

SUMMARY:
Until now, clinicians have been challenged to improve the treatment of biochemically recurrent (BCR) prostate cancer in which prostatic specific antigen (PSA) rises without radiological or clinical progression years after localized treatment (radical prostatectomy or radiation therapy) with or without hormonal treatment. Approximately 50-90% of men with high-risk prostate cancer will experience a BCR. Artesunate has demonstrated anti-tumor activity in both in vivo and in vitro cell lines. It is hypothesized that Artemisia annua (Aa) coffee has the potential to decrease rising PSA among patients with biochemical recurrence of prostate cancer.

DETAILED DESCRIPTION:
This is an open-labeled phase II study of Artemisia annua (Aa) decaf coffee in patients with biochemical recurrence of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Completion of localized therapy (prostatectomy or radiotherapy) for prostate adenocarcinoma (either histologically or cytologically confirmed)
* Biochemical PSA recurrence
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤3
* Total bilirubin ≤ 1.5 x upper normal limit (ULN), and AST (aspartate transaminase) and ALT (alanine transaminase) ≤ 3.0 x ULN
* Patients with a prior or concurrent malignancy (non-prostate) whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as determined by the treating physician are eligible.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any radiological evidence of metastatic disease (determined by standard of care computed tomography (CT) scans of abdomen, pelvis, chest, whole body bone scan or Axium PET/CT scan or prostate specific membrane antigen (PSMA) PET/CT scan).
* Receipt of prior cytotoxic chemotherapy for recurrent prostate cancer
* Use of androgen deprivation therapy (for example, bicalutamide, flutamide, nilutamide, or leuprolide acetate) concurrently or within the previous 3 months.
* Uncontrolled intercurrent illness such as active infections. Other illnesses will be evaluated and eligibility status determined at the discretion of the treating physician and the investigator.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Concomitant use of nevirapine, ritonavir, and strong UGT inducers or strong UGT inhibitors such as phenobarbital, rifampin, carbamazepine, diclofenac, imatinib, axitinib, and vandetanib
* Concurrent use of strong inducers of CYP2A6, including phenobarbital and rifampin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve a 50% decline in PSA levels | 24 weeks
  Proportion of patients who achieve greater than 50% decline in PSA within 24- weeks of coffee treatment.

SECONDARY OUTCOMES:
Change in PSA velocity and slope from pre-treatment to post-treatment | 24 weeks (Baseline and 24 weeks)
  Change in PSA velocity and slope from pre-treatment to post-treatment. Slope and velocity are measured as concentration per unit of time and will have the same units.
Percentage change in serial PSA | 24 weeks (Baseline, 3-mos, 6-mos and post-treatment)
  Percentage change in serial PSA from baseline throughout the treatment period. PSA will be assessed at baseline, 3-mos, 6-mos and at a post-treatment follow-up visit.
Percentage change in serial testosterone levels | 24 weeks (Baseline, 3-mos, 6-mos and post-treatment)
  Percentage change in serial testosterone levels from baseline throughout the treatment period. Testosterone will be assessed at baseline, 3-mos, 6-mos and at a post-treatment follow-up visit.

OTHER OUTCOMES:
Change in plasma concentration of artemisinin and dihydroartemisinin | 24 weeks (Baseline and 24 weeks)
  Changes in plasma concentrations of artemisinin and dihydroartemisinin will be compared pre- and post-treatment with Aa decaf coffee using non-parametric paired test.

CONTACTS AND LOCATIONS:
Overall Officials: Zin Myint, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No